CLINICAL TRIAL: NCT00002349
Title: A Pilot Study to Compare the Antiviral and Immunologic Effects of Stavudine ( d4T ) Versus Placebo in Subjects With Evidence of Recent HIV Infection.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 244A; AI455-029
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2011-04-14 (Estimated); Status verified 2011-04

CONDITIONS: HIV Infections
Keywords: AIDS-Related Complex; Stavudine
MeSH Terms: conditions — HIV Infections; AIDS-Related Complex | interventions — Stavudine

INTERVENTIONS:
Drug: Stavudine

SUMMARY:
To compare the antiviral effect of stavudine ( d4T ) versus placebo in patients with evidence of recent HIV infection.

Also, to compare the immunologic effects and effects on quality of life of d4T in these patients.

DETAILED DESCRIPTION:
Patients receive d4T or placebo every 12 hours for 4 weeks, after which dose decreases (or placebo) every 12 hours. Treatment continues for at least 48 weeks.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Recent HIV infection.
* No prior antiretroviral therapy.
* No acute opportunistic infection at study entry.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Intractable diarrhea.
* Bilateral peripheral neuropathy.
* Any other condition that would preclude study therapy.

Concurrent Medication:

Excluded:

* Myelosuppressive, neurotoxic, or hepatotoxic drugs.

Patients with the following prior condition are excluded:

History of bilateral peripheral neuropathy.

Prior Medication:

Excluded:

* Prior antiretroviral therapy.
* Myelosuppressive, neurotoxic, or cytotoxic agents within 3 months prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 1995-01; Primary Completion 1999-05 (Actual); Study Completion 1999-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - San Diego Naval Hosp, San Diego, California
  - Naval Med Ctr, Portsmouth, Virginia
  - Northwest Med Ctr, Seattle, Washington

REFERENCES:
- [Background] Katlama C, Molina JM, Rozenbaum W, Valantin MA, Modai J, Chauveau E, Ngo Van P, Gres JJ. Stavudine ( D4T ) in HIV infected patients with CD4 less than 350/mm3: results of a double-blind randomized placebo controlled study. Conf Retroviruses Opportunistic Infect. 1996 Jan 28-Feb 1;3rd:89